CLINICAL TRIAL: NCT00219518
Title: Mechano-physiological Approach to Normal Anorectal Function and the Classification of Defecatory Disorders
Brief Title: Mechano-physiological Approach to Anorectal Function
Status: Terminated | Type: Observational
Why Stopped: inadequate no of constip patients
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: American College of Gastroenterology (Other)
Responsible Party: Sponsor
Other Study IDs: HY03-368
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2018-05-25 (Actual); Status verified 2018-05

CONDITIONS: Constipation
Keywords: Defecography; Pelvic floor dyssynergia; Anismus
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

INTERVENTIONS:
Procedure: defecography — insertion of catheter to record pressure. Insertion of barium to outline rectum and fluoroscopy to define change in rectal contour and expulsion of barium during the study.

SUMMARY:
We hypothesize that defecatory disorders can be described in mechanical terms which would allow a mechanistic description of disorders which would in turn allow better directed biofeedback mechanisms to treat disorders of defecation.

DETAILED DESCRIPTION:
Disorders of defecation are very common and the process of defecation remains poorly described. This results in a limited approach to treatment of patients, with limited success. This study will simultaneously measure multiple components of the process of defecation - the abdominal wall and perineal muscle activity, the pressure within the rectum and in the anal canal and the change in shape of the anorectal region of the colon, in order to develop a biomechanical model which can describe the normal and abnormal defecatory process. It is anticipated that, by understanding the process in these terms will allow a new approach to categorizing and describing defecation problems which in turn will lead to more specific approaches of treatment which will be tailored to individual patients. These parameters will compared in volunteers with no defecatory disorders and patients with defecatory disorders who are being referred for defecography as part of their clinical evaluation.

ELIGIBILITY:
Controls

Inclusion Criteria:

* Women
* No defecatory problems
* On no medication which affect bowel habits

Exclusion Criteria:

* Pregnancy

Patients

Inclusion Criteria:

* Difficulty in defecation
* Women

Exclusion criteria:

* Pregnancy
* Medication which can affect bowel movement

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: women with no defecatory dysfunctionl
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2006-02; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
change in shape of anorectum during changes in intraabdominal pressure and defecation | start of anorectal manometry procedure until procedure end
  measure change in dimension over time

CONTACTS AND LOCATIONS:
Overall Officials: Ann Ouyang, MD, Principal Investigator — Penn State College of Medicine and Penn State Milton S. Hershey Medical Center
Locations (1):
- Hershey Medical Center, Hershey, Pennsylvania, United States